CLINICAL TRIAL: NCT04784039
Title: D-Dimer-based Indication for Transesophageal Echocardiography to Exclude Left Atrial Thrombus Before Cardioversion of Non-anticoagulated Atrial Fibrillation: A Multicenter Belgian Study
Acronym: CARDDI-BEL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Principal Investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Version 1.0, 25 February 2021
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEE-group (Active Comparator)
  Interventions: Diagnostic Test: Transesophageal echocardiography
- DD-group (Active Comparator)
  Interventions: Diagnostic Test: D-Dimer analysis

INTERVENTIONS:
Diagnostic Test: Transesophageal echocardiography — Patients randomized to the TEE group will be scheduled for cardioversion with prior TEE
  Arms: TEE-group
Diagnostic Test: D-Dimer analysis — Patients randomized to the DD-group will be scheduled for cardioversion with prior D-Dimer analysis. In case of positive D-Dimer results, TEE will be performed prior to cardioversion
  Arms: DD-group

SUMMARY:
This trial aims at evaluating the number of thromboembolic events post cardioversion in patients receiving a direct current cardioversion with either prior transesophageal echocardiography or D-Dimer (DD) analysis.

Patients in need of a direct current cardioversion (DCCV), meeting the criteria for DCCV with prior transesophageal echocardiography (TEE), will be asked to participate in the CARDDI-BEL study.

Patients will be randomized on a 1:1 ratio to the TEE-group or DD-group. Patients in the TEE-group will receive TEE prior to cardioversion to exclude left atrial thrombus according to current guidelines [1]. In patients randomized to the DD-group, D-Dimer will be analyzed (cut-off defined by DDage). If the DDage > 10x patient's age, the analysis is suggestive for the presence of left atrial thrombus and the cardioversion will be performed with prior TEE. In case of negative DDage, no TEE will be used in the DD-group.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with non-valvular atrial fibrillation scheduled for direct current cardioversion with prior TEE according to current guidelines
* Patients willing to sign informed consent

Exclusion Criteria:

* Cardiac surgery within the previous 90 days.
* Coronary percutaneous transluminal coronary angioplasty/stenting within the previous 90 days or myocardial infarction within the previous 60 days.
* Significant congenital anomaly or other medical problem that in the opinion of the investigator would preclude enrollment
* History of blood clotting disease or bleeding abnormalities.
* Patients with valve implants
* Women who are pregnant
* Aortic aneurysm or dissection
* Documented history of deep vein thrombosis within the last 6 months
* Documented history of pulmonary embolism within the last 6 months
* Unwilling or unable to provide informed consent.
* Recent transient ischemic attack or stroke (90 days)
* Instable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1368 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence in thromboembolic events between both groups after 4 weeks follow-up | up to 4 weeks after cardioversion
  The number of thromboembolic events (stroke, transient ischemic attack, ...) in the TEE and DD-group will be compared

SECONDARY OUTCOMES:
Correlation between D-Dimer-value (ng/L) and number of thrombi visible on TEE | Procedure (At time of cardioversion)
Correlation of DD-value (ng/L) with flow velocity (m/s) in case of spontaneous contrast or suspicion of thrombus in left atrial appendage | Procedure (At time of cardioversion)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan AV